CLINICAL TRIAL: NCT06497257
Title: Effect of Smartphone Overuse on Hand Strength and Function in Physical Therapy Students
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nouran Mohamed Saad, Principal Investigator, Cairo University
Other Study IDs: P.T.REC/012/005125
Record Dates: First submitted 2024-06-29; First posted 2024-07-11 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Smartphone Addiction
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group of high-frequency smartphone users: Male and female subjects, who are high-frequency smartphone users at least for two years before the study.
  Interventions: Other: Evaluating wrist flexor and extensor peak torque; Other: Evaluating functional disability; Other: Evaluating hand grip strength
- Group of low-frequency smartphone users: Male and female subjects, who are low-frequency smartphone users.
  Interventions: Other: Evaluating wrist flexor and extensor peak torque; Other: Evaluating functional disability; Other: Evaluating hand grip strength

INTERVENTIONS:
Other: Evaluating wrist flexor and extensor peak torque — Evaluation of wrist flexor and extensor peak torque
Other: Evaluating functional disability — Evaluation of functional disability
Other: Evaluating hand grip strength — Evaluation of hand grip strength

SUMMARY:
The present study aimed to measure wrist flexor and extensor muscle strength, hand grip strength, wrist pain and function in smartphone addicts and non-addicts

DETAILED DESCRIPTION:
Smartphones have become ubiquitous worldwide, offering significant potential for medical applications by providing healthcare professionals and students with instant access to resources for informed decision-making. However, despite their benefits, overuse of smartphones can lead to physical health issues. Grip strength is recognized as an indicator of overall muscle strength, upper limb function, and various health conditions. Isokinetic testing, a reliable method for measuring muscle performance, has been widely used in studying low back pain but less commonly applied to wrist strength assessment.

Currently, there is a lack of evidence regarding the impact of smartphone overuse on wrist flexor and extensor peak torque, handgrip strength, and function. This research aims to investigate these aspects, providing insights into upper extremity function and potentially aiding ergonomists in addressing musculoskeletal disorders. The study's findings could contribute to the biomechanical evaluation and design of upper extremity tasks, enhance understanding of wrist functioning, and inform ergonomic design considerations. Additionally, the results may help smartphone users adopt better postures and grasping techniques to minimize injuries and maintain hand function, ultimately improving their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age of subjects 18 to 25 years.
* Body mass index from 18, but less than 25 kg/m2.
* Experimental group, healthy subjects who are smartphone users for at least two years prior to study.

Exclusion Criteria:

* Subjects with a history of neurological disorder affecting the upper extremities, vestibular dysfunction, or balance disorder.
* Deformities of elbow or hand.
* Any recent upper limb fracture or trauma.
* Disorders like carpal tunnel syndrome, radiculopathy or tendinopathy.
* Individuals going to the gym or athletes.
* Individuals who smoke.
* Subjects who had cognitive, linguistic or vision impairment which limited their use of instruments and questionnaire.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: They will be selected from the Faculty of Physical Therapy, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Measurement of wrist flexor peak torque | 1 month
  It will be measured by the Biodex system 3 pro isokinetic dynamometer.
Measurement of wrist extensor peak torque | 1 month
  It will be measured by the Biodex system 3 pro isokinetic dynamometer.
Assessment of functional disability | 1 month
  It will be assessed by the patient-related wrist and hand evaluation (PRWHE) questionnaire.
Measurement of hand grip strength | 1 month
  It will be measured by a JAMAR Handheld Dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa Kenawy, PhD, Study Chair — Faculty of physical therapy, Cairo University, Giza, Egypt.
Locations (1):
- Nouran Mohamed Saad, Cairo, Egypt